CLINICAL TRIAL: NCT03928405
Title: The Effect of Virtual Reality Application on Balance and Gait Speed in Individuals With Alzheimer's Dementia
Brief Title: Effect of Virtual Reality on Balance and Gait Speed With Alzheimer's Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meral SERTEL, Assoc. Prof., Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alzheimer,Virtual Reality
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer's Dementia
Keywords: Alzheimer's Dementia; Balance; Gait Speed; Virtual Reality
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study consisted of 32 subjects, which were diagnosed as mild or moderate AD by the neurologist. The balance, fall risks and gait speed were assessed. Training group was trained with games selected from different categories such as balance and aerobic exercises with Nintendo Wii virtual reality device for 6 weeks, 1 session 30 min, 2 times a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): The subjects were evaluated with the case report form, the balance and fall risks, the Tinetti Gait and Balance Test (TGBT) and the 5-times Sit to Stand Test, while the gait speed was assessed by the Gait Speed Measurement Test (GSMT). The virtual reality group was trained with games selected from different categories such as balance and aerobic exercises with Nintendo Wii virtual reality device for 6 weeks, 1 session 30 min, 2 times a week. In the control group, no treatment was performed during this period and routine medical treatments were continued. In the first session, each Nintendo Wii components were introduced to each individual. The selected games and how they were played were taught to each individual by the physiotherapist and practically taught. The games were played with the help of physiotherapists in the first session so that individuals could transfer the correct weight on the Nintendo Wii balance board and to use the game console's control.
  Interventions: Other: Exercises with Nintendo Wii virtual reality device
- Control Group (No Intervention): The sociodemographic characteristics of the subjects were evaluated with the case report form, the balance and fall risks, the Tinetti Gait and Balance Test (TGBT) and the 5-times Sit to Stand Test, while the gait speed was assessed by the Gait Speed Measurement Test (GSMT).the control group was reevaluated at the end of the 6th week after the initial evaluation. After the study was completed, training was given to the volunteers from the control group.

INTERVENTIONS:
Other: Exercises with Nintendo Wii virtual reality device — In the first session, each Nintendo Wii components were introduced to each individual. The selected games and how they were played were taught to each individual by the physiotherapist and practically taught. The games were played with the help of physiotherapists in the first session so that individuals could transfer the correct weight on the Nintendo Wii balance board and to use the game console's control. The patient was supported with verbal and physical feedback when the patient played incorrectly during the games in the next sessions. Games that require serious balance and coordination were considered as a difficult activity for the patient and were not used in this study. The difficulty of the games was set to the simplest level for each patient. As the patients were successful the games' difficulty level was upgraded. The difficulty of the games has been increased according to the classification determined by the Nintendo Wii device.
  Other Names: Virtual reality game
  Arms: Virtual reality group

SUMMARY:
The aim of study is to investigate the effect of virtual reality application on balance and gait speed in individuals with Alzheimer's Dementia.

DETAILED DESCRIPTION:
The aim of study is to investigate the effect of virtual reality application on balance and gait speed in individuals with Alzheimer's Dementia. The study consisted of 32 subjects, which were diagnosed as mild or moderate AD by the neurologist. The balance, fall risks and gait speed were assessed. Training group was trained with games selected from different categories such as balance and aerobic exercises with Nintendo Wii virtual reality device for 6 weeks, 1 session 30 min, 2 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Having mild or moderate severity of AD
* Lack of communication difficulties or problems
* Volunteering to participate in the study
* Cerebrovascular event,
* Having disturbing the balance and coordination of neurological disease such as Parkinson, MS,
* Mini Mental Test Score, 18 to 24 points from being scored
* being 65-80 aged.

Exclusion Criteria:

* Patients diagnosed with dementia (infection, vascular, hematological diseases), patients who could not be contacted during the follow-up period or who did not come to control, cardiac and cerebrovascular event,
* Endocrine disorder, fluid-electrolyte imbalance and infection
* Patients with malignancy and malignancy, chemotherapy and radiotherapy,
* Patients with delirium or depression
* Those with protective sensation loss (those with Semmes-Weinstein Monofilament Thickness 4.56 and above)
* patients with lower or upper extremity amputations at any level

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
The Tinetti Gait and Balance Test (TGBT) | 15 minute
  TGBT consists of balance and gait subheadings. For balance, there are 13 items, and 9 items for gait. Items are scored as 0 (abnormal), 1 (adaptive) and 2 (normal) for balance, 0 (abnormal), 1 (normal) for gait. The maximum balance score of the patient is 26 and the maximum gait score is 9. Total score (balance + walking) is 35 points.
The 5-times Sit to Stand Test | 1 minute
  5 times sit to stand test is a test that evaluates the functional strength of the lower extremity, balance and fall risk. In order to perform this test, a standard size chair with a stopwatch and a flat back is required. We said to the patient that "Please cross your arms to the other shoulder, and when I say start, sit and stand 5 times in the fastest and straightest way you can". I will measure your time with the stopwatch. The rank of the patients was told to them for sit and stand. In the elderly, if the duration of this period is more than 12 seconds indicated the risk of falling, if it is over 15 seconds, this is an indicator of the presence of a risk of repetitive drop
The Gait Speed Measurement Test (GSMT) | 5 minute
  For GSMT, individuals were asked to walk at a speed they wanted on a flat surface of 14 m. Signs were placed on the 2nd and 12th meters of the test area to minimize the speed changes between walking start and walking finish, and to make a more objective measurement. The walking time at this 10-meter distance was measured with the stopwatch and the results were recorded in sec and the walking speed was determined
Mini Mental State Test | 15 minute
  It was used to determine the cognitive state before the training. The Mini-Mental State Test was first published by Folstein et al. It consists of eleven items under 5 main headings: orientation, record memory, attention and calculation, recall and language, and the total score is evaluated over 30 points.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma KABAKCI, Study Chair — Karaman Ahmet Mete Nursing Home for the Elderly Care
Locations (2):
- Turkey (Türkiye) (2):
  - Kirikkale University, Kırıkkale, Fabrikalar Street
  - Kirikkale Universtiy, Kırıkkale, Fabrikalar Street

IPD SHARING:
Plan to Share IPD: No